CLINICAL TRIAL: NCT04059549
Title: Building and Pilot Testing a Couples-based Smartphone Systems to Address Alcohol Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: University of Massachusetts, Worcester (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-0696; A195010 (Other: UW Madison); ENGR/INDUSTRIAL ENGR (Other: UW Madison); 1R34AA025675-01A1 (NIH); Protocol Version 7/6/2020 (Other: UW Madison)
Record Dates: First submitted 2019-08-14; First posted 2019-08-16 (Actual); Results first posted 2022-12-07 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2022-11

CONDITIONS: Alcohol Use Disorder; Couples; Behavior, Addictive
MeSH Terms: conditions — Alcoholism; Behavior, Addictive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A-CHESS Drinker (Active Comparator): Patients randomized to the A-CHESS group will receive the A-CHESS app on a smartphone.
  Interventions: Behavioral: A-CHESS
- PartnerCHESS Drinker (Experimental): Patients randomized to the PartnerCHESS group will receive all A-CHESS services listed above, plus learning modules and resources from Alcohol-based Couple Therapy.
  Interventions: Behavioral: PartnerCHESS
- A-CHESS Partner (Active Comparator): Patient's partner randomized to the A-CHESS group will receive the A-CHESS app on a smartphone.
  Interventions: Behavioral: A-CHESS
- PartnerCHESS Partner (Experimental): Patient's partner randomized to the PartnerCHESS group will receive all A-CHESS services listed above, plus learning modules and resources from Alcohol-based Couple Therapy.
  Interventions: Behavioral: PartnerCHESS

INTERVENTIONS:
Behavioral: PartnerCHESS — Patients randomized to the PartnerCHESS group will receive all A-CHESS services plus the following services from ABCT:
  Urge discussion. Daily EMAs will track preconditions for relapse (urges), review urge reduction options on PartnerCHESS, and encourage discussions between partners on the causes of and ways to reduce urges.
  Homework checklist. Tracks which interventions the couple is using/practicing, along with resources to help.
  Relapse plan. Monitoring and reminders of steps planned for relapse prevention. Reminders. Reminders to notice something positive in partner, of reasons to stay sober, to take meds, etc.
  Trigger identification and removal. During set-up, patient and partner enter triggers. PartnerCHESS will quiz couples on upcoming trigger events and remind them of ways to address each.
  Arms: PartnerCHESS Drinker; PartnerCHESS Partner
Behavioral: A-CHESS — A-CHESS control group
  Arms: A-CHESS Drinker; A-CHESS Partner

SUMMARY:
This project will develop and pilot test a new smartphone-based system for AUD patients, their partners, and clinicians called PartnerCHESS. PartnerCHESS will integrate key features of ABCT and A-CHESS. PartnerCHESS will also include a Clinician Report to automatically alert clinicians of patients at risk of relapse and offer other information on how recovery is proceeding. The project has three specific aims:

1. Integrate A-CHESS with key features of ABCT to create PartnerCHESS to serve patients, partners, and clinicians.
2. Conduct a pilot test (a small randomized clinical trial) of PartnerCHESS to estimate effect size and refine the protocol, procedures, recruitment strategy, measurements, and operations for use in a large RCT.

3a. Decide whether to pursue an R01 application, and if so, 3b. plan for the R01.

DETAILED DESCRIPTION:
Alcohol use disorder (AUD) is one of the most common substance use disorders. Yet only a small fraction of people who need treatment receive it, and most of them get only short-term support even though continuing care has been shown to be much more effective. Partner support can be critical to recovery, but many partners do not know how to support their partners' recovery or manage their own responses to it. Clinicians also lack evidence of the efforts patients are making toward recovery. Treating couples in which one member is recovering from AUD has been shown to be efficacious; in particular, Alcohol Behavioral Couples Therapy (ABCT) has shown positive outcomes. Still, ABCT has not been widely adopted, in part because of practical problems such as the stigma that goes with the partner needing to go to an addiction treatment agency to participate. A-CHESS is a smartphone-based system proven to substantially reduce relapse rates, but A-CHESS serves only the patient.

This project will develop and pilot test a new smartphone-based system for AUD patients, their partners, and clinicians called PartnerCHESS. PartnerCHESS will integrate key features of ABCT and A-CHESS. PartnerCHESS will also include a Clinician Report to automatically alert clinicians of patients at risk of relapse and offer other information on how recovery is proceeding. The project has three specific aims:

1. Integrate A-CHESS with key features of ABCT to create PartnerCHESS to serve patients, partners, and clinicians.
2. Conduct a pilot test (a small randomized clinical trial) of PartnerCHESS to estimate effect size and refine the protocol, procedures, recruitment strategy, measurements, and operations for use in a large RCT.

3a. Decide whether to pursue an R01 application, and if so, 3b. plan for the R01.

The project would engage 6 couples to help design PartnerCHESS, test its usability and give feedback on its utility. Once ready, the system would be tested by 34 other couples randomized to receive either PartnerCHESS + treatment as usual (TAU) or A-CHESS + TAU for a 6-month trial. The investigators will collect survey data at baseline, 2, 4, and 6 months and analyze it to see if a large clinical trial holds promise and, if so, produce an application to support a full-scale trial based on the technology developed and the research procedures employed in the pilot test.

The study is important to public health because of the scope of the alcohol abuse and the potential of technology to improve the lives of both patients and partners. If successful, such technology could greatly broaden the reach and impact of AUD treatment in general and couples therapy in particular.

ELIGIBILITY:
A total of 34 dyads were recruited.

Patients and partners:

* Must be 18 or older
* Not have a mental or physical condition that limits smartphone use
* Cannot have experienced serious Interpersonal Violence Intimate Partner Violence (IPV) in the index (therapy) relationship in the past year
* Not have a history of schizophrenia

Patients:

* Must have a DSM-5 diagnosis of alcohol use disorder or meet NIAAA guidelines for risky drinking.
* Have had at least one alcoholic drink in the last 6 months

Partners:

* Must be a spouse, or in a 6-month or longer committed romantic relationship
* Willing to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2021-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David H Gustafson, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- Stanley Street Treatment and Resources, Fall River, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gustafson DH Sr, Gustafson DH Jr, Mares ML, Johnston DC, Vjorn OJ, Curtin JJ, Epstein EE, Bailey GL. Couple-Focused Smartphone Intervention to Reduce Problem Drinking: Pilot Randomized Control Trial. JMIR Form Res. 2024 Nov 1;8:e58622. doi: 10.2196/58622. PMID 39486022

RESULTS

PARTICIPANT FLOW:
Groups:
- A-CHESS Dyads: Patients randomized to the A-CHESS group will receive the A-CHESS app on a smartphone.
  A-CHESS: A-CHESS control group
- PartnerCHESS Dyads: Patients randomized to the PartnerCHESS group will receive all A-CHESS services listed above, plus learning modules and resources from Alcohol-based Couple Therapy.
  PartnerCHESS: Patients randomized to the PartnerCHESS group will receive all A-CHESS services plus the following services from ABCT:
  Urge discussion. Daily EMAs will track preconditions for relapse (urges), review urge reduction options on PartnerCHESS, and encourage discussions between partners on the causes of and ways to reduce urges.
  Homework checklist. Tracks which interventions the couple is using/practicing, along with resources to help.
  Relapse plan. Monitoring and reminders of steps planned for relapse prevention. Reminders. Reminders to notice something positive in partner, of reasons to stay sober, to take meds, etc.
  Trigger identification and removal. During set-up, patient and partner enter triggers. PartnerCHESS will quiz couples on upcoming trigger events and remind them of ways to address each.
Period: Overall Study
Arm/Group | A-CHESS Dyads | PartnerCHESS Dyads
Started | 32 (16 dyads) | 36 (18 dyads)
Completed | 30 (15 dyads) | 36 (18 dyads)
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- PartnerCHESS Drinker: Patients randomized to the PartnerCHESS group will receive all A-CHESS services listed above, plus learning modules and resources from Alcohol-based Couple Therapy.
  PartnerCHESS: Patients randomized to the PartnerCHESS group will receive all A-CHESS services plus the following services from ABCT:
  Urge discussion. Daily EMAs will track preconditions for relapse (urges), review urge reduction options on PartnerCHESS, and encourage discussions between partners on the causes of and ways to reduce urges.
  Homework checklist. Tracks which interventions the couple is using/practicing, along with resources to help.
  Relapse plan. Monitoring and reminders of steps planned for relapse prevention. Reminders. Reminders to notice something positive in partner, of reasons to stay sober, to take meds, etc.
  Trigger identification and removal. During set-up, patient and partner enter triggers. PartnerCHESS will quiz couples on upcoming trigger events and remind them of ways to address each.
- A-CHESS Partner: Participants randomized to the A-CHESS group will receive the A-CHESS app on a smartphone.
  A-CHESS: A-CHESS control group
- PartnerCHESS Partner: Participants randomized to the PartnerCHESS group will receive all A-CHESS services listed above, plus learning modules and resources from Alcohol-based Couple Therapy.
  PartnerCHESS: Patients randomized to the PartnerCHESS group will receive all A-CHESS services plus the following services from ABCT:
  Urge discussion. Daily EMAs will track preconditions for relapse (urges), review urge reduction options on PartnerCHESS, and encourage discussions between partners on the causes of and ways to reduce urges.
  Homework checklist. Tracks which interventions the couple is using/practicing, along with resources to help.
  Relapse plan. Monitoring and reminders of steps planned for relapse prevention. Reminders. Reminders to notice something positive in partner, of reasons to stay sober, to take meds, etc.
  Trigger identification and removal. During set-up, patient and partner enter triggers. PartnerCHESS will quiz couples on upcoming trigger events and remind them of ways to address each.
- Total: Total of all reporting groups
Arm/Group | A-CHESS Drinker | PartnerCHESS Drinker | A-CHESS Partner | PartnerCHESS Partner | Total
Number analyzed (Participants) | 15 | 18 | 15 | 18 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.33 (12.43) | 37.83 (10.53) | 40.93 (12.40) | 38.50 (10.27) | 39.97 (11.30)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 3 | 4 | 13 | 13 | 33
  Male | 12 | 13 | 2 | 5 | 32
  Prefer not to say | 0 | 1 | 0 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 0 | 0 | 3
  Not Hispanic or Latino | 13 | 17 | 15 | 18 | 63
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 0 | 3 | 6
  White | 12 | 14 | 12 | 15 | 53
  More than one race | 2 | 2 | 2 | 0 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Living with partner [Count of Participants; unit: Participants] | 12 | 15 | 12 | 16 | 55
Alcohol use disorder severity (DSM-5) [Count of Participants; unit: Participants] — This was not measured for partners, because they are not being assessed for Alcohol use disorder. Population: The number analyzed differs from overall number because partners were not being assessed for Alcohol use disorder.
  Participants
    number analyzed (Participants) | 15 | 18 | 0 | 0 | 33
    Mild 2-3 | 1 | 0 | 0 | 0 | 1
    Moderate 4-5 | 2 | 0 | 0 | 0 | 2
    Severe 6+ | 12 | 18 | 0 | 0 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With no Heavy Drinking
Description: At each time of measurement, a timeline follow-back interview was conducted for the past 60 days. Risky drinking day was be defined as greater than 4 drinks for men and greater than 3 drinks for women in 2 hours.
Time Frame: baseline, 2, 4, and 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | A-CHESS Drinker | PartnerCHESS Drinker
Number analyzed (Participants) | 15 | 18
Participants
  Baseline | 1 | 2
  2 months | 1 | 5
  4 months | 5 | 10
  6 months | 6 | 13

2. Primary Outcome: Percentage of Days With Heavy Drinking
Description: At each time of measurement, a timeline follow-back interview was conducted for the past 60 days.
Time Frame: baseline, 2, 4, and 6 months
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | A-CHESS Drinker | PartnerCHESS Drinker
Number analyzed (Participants) | 15 | 18
percentage of days
  Baseline | 51.7 (38.4) | 50.3 (34.7)
  2 months | 46.7 (39.4) | 28.6 (28.0)
  4 months | 34.9 (40.5) | 18.2 (29.2)
  6 months | 37.4 (44.6) | 17.7 (31.7)

3. Primary Outcome: Percentage of Days With Any Drinking
Description: At each time of measurement, a timeline follow-back interview was conducted for the past 60 days.
Time Frame: Baseline, 2, 4, 6 months
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | A-CHESS Drinker | PartnerCHESS Drinker
Number analyzed (Participants) | 15 | 18
percentage of days
  Baseline | 72.8 (33.5) | 73.6 (30.0)
  2 months | 58.3 (38.9) | 59.6 (36.2)
  4 months | 48.3 (42.3) | 46.6 (44.7)
  6 months | 52.7 (43.5) | 48.4 (44.5)

4. Secondary Outcome: Psychological Distress
Description: Drinkers' and partners' psychological distress was assessed by the OQ-45 scale. Response options range from 0-4, with items 1, 12, 13, 20, 21, 24, 31, 37, and 43 reversed; items are summed (i.e., a possible range of 0-180). High scores suggest distress (anxiety, depression, somatic problems, stress), difficulties in interpersonal relationships and social roles (e.g., work), and low quality of life, with scores of 63 or more indicating symptoms of clinical significance, and changes of 14 points or more considered reliable.
Time Frame: baseline, 2, 4, and 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- PartnerCHESS Partner: Patient's partner randomized to the PartnerCHESS group will receive all A-CHESS services listed above, plus learning modules and resources from Alcohol-based Couple Therapy.
  PartnerCHESS: Patients randomized to the PartnerCHESS group will receive all A-CHESS services plus the following services from ABCT:
  Urge discussion. Daily EMAs will track preconditions for relapse (urges), review urge reduction options on PartnerCHESS, and encourage discussions between partners on the causes of and ways to reduce urges.
  Homework checklist. Tracks which interventions the couple is using/practicing, along with resources to help.
  Relapse plan. Monitoring and reminders of steps planned for relapse prevention. Reminders. Reminders to notice something positive in partner, of reasons to stay sober, to take meds, etc.
  Trigger identification and removal. During set-up, patient and partner enter triggers. PartnerCHESS will quiz couples on upcoming trigger events and remind them of ways to address each.
Arm/Group | A-CHESS Drinker | PartnerCHESS Drinker | A-CHESS Partner | PartnerCHESS Partner
Number analyzed (Participants) | 15 | 18 | 15 | 18
score on a scale
  Baseline | 54.5 (31.1) | 66.3 (27.4) | 44.5 (23.4) | 53.6 (21.8)
  2 months | 51.7 (29.5) | 65.7 (28.2) | 46.8 (24.1) | 53.0 (20.8)
  4 months | 40.3 (25.0) | 59.7 (27.4) | 41.5 (16.1) | 52.9 (27.3)
  6 months | 48.8 (25.3) | 52.1 (25.8) | 43.2 (25.4) | 54.8 (29.1)

5. Secondary Outcome: Relationship Satisfaction
Description: Drinkers' and partners' relationship satisfaction was assessed by the Dyadic Adjustment Scale-Brief (DAS-7) plus item 32 from the DAS-32. Response options ranged 0-5 on most items and 0-6 on item 7 of the DAS-7 (possible scores range from 0 to 41). Consistent with scoring instructions for the DAS-7, items were summed, with higher scores indicating more satisfaction.
Time Frame: baseline, 2, 4, and 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | A-CHESS Drinker | PartnerCHESS Drinker | A-CHESS Partner | PartnerCHESS Partner
Number analyzed (Participants) | 15 | 18 | 15 | 18
score on a scale
  Baseline | 28.4 (4.1) | 27.5 (7.3) | 27.4 (6.8) | 27.6 (6.4)
  2 months | 27.9 (4.3) | 27.0 (8.1) | 26.9 (6.5) | 26.5 (7.7)
  4 months | 30.0 (4.4) | 28.1 (7.7) | 27.1 (6.2) | 25.4 (6.7)
  6 months | 29.4 (5.9) | 27.4 (7.9) | 27.5 (6.6) | 24.3 (7.3)

6. Secondary Outcome: Perceptions of Family Environment - Cohesion
Description: Drinkers and partners both completed the 9-item Cohesion and 9-item Conflict scales from the Family Environment Scale. Responses were true/false statements, with higher scores indicating more cohesion or conflict. Possible scores range from 4 to 65.
Time Frame: Baseline, 2, 4, 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | A-CHESS Drinker | PartnerCHESS Drinker | A-CHESS Partner | PartnerCHESS Partner
Number analyzed (Participants) | 15 | 18 | 15 | 18
score on a scale
  Baseline | 54.9 (11.8) | 52.6 (9.9) | 52.6 (10.5) | 47.4 (15.8)
  2 months | 53.2 (10.4) | 50.4 (13.5) | 52.3 (12.6) | 50.7 (13.4)
  4 months | 58.6 (8.0) | 54.8 (14.6) | 56.4 (11.8) | 55.2 (9.9)
  6 months | 57.3 (8.6) | 54.8 (15.9) | 57.2 (12.8) | 50.7 (17.4)

7. Secondary Outcome: Perceptions of Family Environment - Conflict
Description: Drinkers and partners both completed the 9-item Cohesion and 9-item Conflict scales from the Family Environment Scale. Responses were true/false statements, with higher scores indicating more cohesion or conflict. Possible scores range from 33 to 80.
Time Frame: Baseline, 2, 4, 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | A-CHESS Drinker | PartnerCHESS Drinker | A-CHESS Partner | PartnerCHESS Partner
Number analyzed (Participants) | 15 | 18 | 15 | 18
score on a scale
  Baseline | 46.2 (14.2) | 48.6 (12.7) | 47.1 (12.4) | 52.8 (13.1)
  2 months | 40.6 (12.3) | 45.3 (11.3) | 45.7 (11.0) | 45.4 (11.3)
  4 months | 40.6 (9.8) | 43.4 (11.7) | 43.8 (10.6) | 43.2 (10.5)
  6 months | 42.3 (13.2) | 43.6 (10.5) | 43.1 (8.7) | 46.7 (12.7)

8. Secondary Outcome: Commitment to Sobriety
Description: Drinkers completed the 5-item Commitment to Sobriety Scale. Response options ranged 1-5 for a total possible range of scores from 5-25; with higher scores suggesting more commitment.
Time Frame: Baseline, 2, 4, 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | A-CHESS Drinker | PartnerCHESS Drinker
Number analyzed (Participants) | 15 | 18
score on a scale
  Baseline | 16.2 (6.4) | 15.9 (4.7)
  2 months | 15.2 (4.6) | 15.1 (6.2)
  4 months | 15.7 (6.1) | 17.8 (4.7)
  6 months | 15.9 (6.9) | 17.4 (5.7)

9. Secondary Outcome: Peer Support
Description: Partners reported on the availability of peer support using the 5-item McTavish Bonding Scale. Response options ranged 1-5 for a total possible range of scores from 5-25; with higher scores suggesting more support.
Time Frame: Baseline, 2, 4, 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | A-CHESS Partner | PartnerCHESS Partner
Number analyzed (Participants) | 15 | 18
score on a scale
  Baseline | 13.4 (6.4) | 10.8 (4.2)
  2 months | 13.1 (7.5) | 16.1 (3.8)
  4 months | 11.5 (4.8) | 14.8 (3.9)
  6 months | 12.9 (5.7) | 15.6 (5.2)

ADVERSE EVENTS:
Time Frame: Up to 6 months
Groups:
- A-CHESS: Patients randomized to the A-CHESS group will receive the A-CHESS app on a smartphone.
  A-CHESS: A-CHESS control group
- PartnerCHESS: Patients randomized to the PartnerCHESS group will receive all A-CHESS services listed above, plus learning modules and resources from Alcohol-based Couple Therapy.
  PartnerCHESS: Patients randomized to the PartnerCHESS group will receive all A-CHESS services plus the following services from ABCT:
  Urge discussion. Daily EMAs will track preconditions for relapse (urges), review urge reduction options on PartnerCHESS, and encourage discussions between partners on the causes of and ways to reduce urges.
  Homework checklist. Tracks which interventions the couple is using/practicing, along with resources to help.
  Relapse plan. Monitoring and reminders of steps planned for relapse prevention. Reminders. Reminders to notice something positive in partner, of reasons to stay sober, to take meds, etc.
  Trigger identification and removal. During set-up, patient and partner enter triggers. PartnerCHESS will quiz couples on upcoming trigger events and remind them of ways to address each.
Arm/Group | A-CHESS | PartnerCHESS
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/36
Other Adverse Events (participants affected / at risk) | 0/30 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-20): https://cdn.clinicaltrials.gov/large-docs/49/NCT04059549/Prot_SAP_000.pdf